CLINICAL TRIAL: NCT02142036
Title: N-of-1 Trial of Actionable Target Identification in Metastatic Cancer for Palliative Systemic Therapy
Brief Title: N-of-1 Trial: Actionable Target Identification in Metastatic Cancer for Palliative Systemic Therapy
Acronym: MetAction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kjersti Flatmark, National coordinator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MetAction
Record Dates: First submitted 2014-04-13; First posted 2014-05-20 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Cancer
Keywords: Metastatic disease; Metastasis; Targeted therapy; Solid tumor; Personalized medicine; N-of-1 trial
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cetuximab; Panitumumab; Gefitinib; Erlotinib Hydrochloride; Crizotinib; Trastuzumab; Lapatinib; Imatinib Mesylate; Dasatinib; nilotinib; Vemurafenib; Everolimus; temsirolimus; Sunitinib; ruxolitinib; vandetanib; Afatinib; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATI based targeted therapy. (Experimental): EMA-approved ATI based targeted therapy. Patients will receive therapy based on molecular aberrations identified in the metastatic lesion.
  Interventions: Drug: EMA-approved ATI based targeted therapy

INTERVENTIONS:
Drug: EMA-approved ATI based targeted therapy — All drugs that may be used in the study are approved by EMA for treatment of disseminated cancer in the palliative setting, but not for the particular tumor type in question.
  Other Names: Cetuximab; Panitumumab; Gefitinib; Erlotinib; Crizotinib; Trastuzumab; Lapatinib; Imatinib; Dasatinib; Nilotinib; Vemurafenib; Everolimus; Temsirolimus; Sunitinib; Ruxolitinib; Vandetanib.; Afatinib; Dabrafenib

SUMMARY:
The metastatic lesions may be very different from the primary tumor because of intrinsic tumor heterogenity, clonal selection through metastatic process and following previous cytotoxic treatments. Metastatic tumor harboring actionable targets or signaling pathways may respond to inhibitory agents directed against specific aberrations irrespective of tumor origin. In the MetAction study, patients will receive therapy based on molecular aberrations in the metastatic lesions, actionable target identification (ATI), rather than on histological tumor type.

The ATI rate in an unselected metastatic patient population is uncertain, and response rates associated with ATI based targeted therapy have hardly been reported. In this perspective, The MetAction study is essentially a feasibility study aiming to tailor metastatic cancer therapy based on genomic profiles.

DETAILED DESCRIPTION:
Recognizing the rapidly increasing number of drugs targeting specific molecular aberrations in cancer, it is necessary to define rational strategies to make such treatment available to Norwegian cancer patients.These targeted drugs are extremely costly and have significant side effects, although presumably to a lesser extent than many of the classic cytotoxic drugs available. Thus, in the interest of the patient in question and the society in general, it is important to give the right drug to the right patient and to the presumably right time in the disease course.

Hitherto, most of the drugs in question are given in the palliative setting, i.e. to patients with disseminated metastatic disease. The metastatic lesion may be very different from the primary tumor, and hence, it is rational to analyze the tumor to be treated, the metastatic lesion(s), for the presence of molecular aberrations, rather than basing treatment decisions on molecular features known to be present in a particular tumor type or in the primary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer and progression by RECIST 1.0 evaluated by internal review on at least one prior regimen of established palliative systemic therapies for advanced disease and eligibility for repeat biopsy sampling. The patient must have received ≥6 weeks of the previous treatment. Only patients who have no other standard treatment option or were the treatment option is considered to offer the patients only minor benefit may be included in the study.
* Radiological evaluation intervals on last prior therapy (period A) must have been 6 to 12 weeks.
* At least one measurable lesions (>10mm on CT-scan) according to RECIST 1.0.
* Age ≥ 18 years. Eastern Cooperative Oncology Group (ECOG) performance status 1 or lower.
* Life expectancy of more than 3 months.
* Adequate bone marrow function without current use of colony-stimulating factors: Neutrophils ≥1.5 x109/l; Platelets ≥100 x109/l; Hb >10 g/dl, INR within normal level.
* Adequate liver function: AST/ALT ≤5x ULN; Bilirubin ≤2x ULN, albumin >30 g/l.
* Adequate renal function: Creatinine ≤1.5x ULN.
* Be able to use recommended dose of the selected targeted therapy as described in the drug specific SPC.
* Be able to comply with the protocol.
* Fertile men and women must be willing to use effective contraceptives.
* Provide written (signed) informed consent to participate in the trial prior to any trial specific screening procedures.

Exclusion Criteria:

* Metastatic disease from more than one malignancy.
* Untreated or symptomatic brain metastasis (patients must be symptom-free without the use of corticosteroids).
* Any reason why, in the opinion of the investigator, the patient should not participate.
* Pregnancy.
* Breastfeeding
* Anticoagulation with coumarin derivatives.
* Radiation therapy within 4 weeks of start of treatment.
* Need to use medications contraindicated according to SPC of the different drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of initiation of study treatment until the date of first documented progression or date of death, from any cause, whichever came first, assessed up to 24 months.
  Comparing the PFS using therapy selected by ATI in a patient's tumor (period B) with the PFS for the most recent therapy on which the patient had just experienced progression (period A). The ATI-selected therapy is defined as having benefit for the patient if PFS period B/PFS in period A ratio is ≥ 1.3.

SECONDARY OUTCOMES:
Overall response rate (ORR) | From date of initiation of study treatment until the date of first documented progression, assessed up to 24 months.
  The sum of partial responses (PS) plus complete responses (CR).
Overall survival (OS) | From date of initiation of study treatment until date of death, from any cause, assessed up to 24 months.

OTHER OUTCOMES:
Overall clinical benefit rate (ORR + stable disease [SD] ≥ 6 months) | From date of initial response to date of first documented progression, assessed up to 24 months.
ATI rate | From date of screening of first included patient until date of completion of screening phase, an expected time period of 24 months..
PFS in ATI lesions only. | From date of initiation of study treatment until date of first documented progression in ATI lesions, assessed up to 24 months.
Health Related Quality of Life (HRQoL) Questionnaire | From date of initiation of study treatment until date of end of study visit, an expected average of 4 months.
  Assessed by the subject questionnaire EORTC Quality of Life Questionnaire Core 30 (QlQ-C30) at baseline, every 8 week during treatment and at end of study visit.
Toxicity grade 3-5 | From date of initiation of study treatment until date of follow-up visit, an expected average of 5 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Flatmark, MD PhD, Study Chair — Oslo University Hospital; Svein Dueland, MD, Principal Investigator — Oslo University Hospital; Anne Hansen Ree, Prof. MD PhD, Principal Investigator — University Hospital, Akershus
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lillestrøm
  - The Norwegian Radium Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ree AH, Maelandsmo GM, Flatmark K, Russnes HG, Gomez Castaneda M, Aas E. Cost-effectiveness of molecularly matched off-label therapies for end-stage cancer - the MetAction precision medicine study. Acta Oncol. 2022 Aug;61(8):955-962. doi: 10.1080/0284186X.2022.2098053. Epub 2022 Aug 9. PMID 35943168
- [Derived] Ree AH, Nygaard V, Boye K, Heinrich D, Dueland S, Bergheim IR, Johansen C, Beiske K, Negard A, Lund-Iversen M, Nygaard V, Hovig E, Nakken S, Nasser S, Julsrud L, Reisse CH, Ruud EA, Kristensen VN, Florenes VA, Geitvik GA, Lingjaerde OC, Borresen-Dale AL, Russnes HG, Maelandsmo GM, Flatmark K. Molecularly matched therapy in the context of sensitivity, resistance, and safety; patient outcomes in end-stage cancer - the MetAction study. Acta Oncol. 2020 Jul;59(7):733-740. doi: 10.1080/0284186X.2020.1742377. Epub 2020 Mar 25. PMID 32208873